CLINICAL TRIAL: NCT04659291
Title: Prospective Study on Patients With Obstructive Sleep Apnea in Hong Kong (PrOSA)
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Susanna SS Ng, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: PrOSA study/2020
Record Dates: First submitted 2020-08-31; First posted 2020-12-09 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: cognitive function
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is a common disorder with prevalence rates of at least 4% among the middle-aged male Caucasians and Hong Kong (HK) Chinese populations. It is characterized by repetitive episodes of upper airway obstruction, causing intermittent hypoxia, sleep fragmentation, disabling daytime sleepiness, impaired cognitive function and poor health status. OSAS patients are at increased risks of non-fatal and fatal cardiovascular morbidity and mortality including sudden death, in addition to being more prone to road traffic accidents. However, there is no long term follow up of patients with OSAS on the incidence of cardiovascular disease, compliance on the therapy and the impact of the quality of life. The study is aimed to carry out a prospective observational study assessing the role of OSAS as a possible cause of increased cardiovascular risk and cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* suspected obstructive sleep apnea syndrome
* aged 18 or above
* must be able to speak, read and understand Chinese or English
* possess the ability to respond to questions and follow instructions.

Exclusion Criteria:

* already treated sleep apnea,
* a limited life expectancy due to illness unrelated to sleep apnea
* human immunodeficiency virus (HIV),
* advanced renal disease,
* uncontrolled malignancies
* documented alcohol or drug abuse up to 1 year prior to inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients are recruited from the Respiratory Clinic at the Prince of Wales Hospital with clinical suspicion of sleep-disordered breathing. The Respiratory Clinic receives referral from hospital specialists and general practitioners. The clinical evaluation procedure includes an interview by a respiratory specialist followed by either an inpatient polysomnography or home polygraphic study according to the patients' clinical characteristics and preference in concordance of the guidelines from the American Academy of Sleep Medicine (AASM). Sleep records will be scored based on standardized criteria of AASM.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2028-08-29 (Estimated); Study Completion 2028-08-29 (Estimated)

PRIMARY OUTCOMES:
incidence of Cardiovascular disease | 5 years

SECONDARY OUTCOMES:
Change of Montreal Cognitive Assessment score (MoCA) | 5 years
  MoCA scores range between 0 and 30. Higher scores mean a better cognitive function.
Change of Epworth Sleepiness Score | 5 years
  The Epworth Sleepiness Scale can be used to assess daytime sleepiness. The scores range between 0 and 24. Higher scores mean more sleepiness.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong, Hong Kong, Please Select, Hong Kong

IPD SHARING:
Plan to Share IPD: No